CLINICAL TRIAL: NCT01573637
Title: Six Month, Double Blind, Placebo-controlled Trial of the Efficacy of Raloxifene as an Adjuvant Treatment of the Negative Symptoms of Schizophrenia in Post-menopausal Women
Brief Title: Raloxifene as an Adjuvant Treatment of the Negative Symptoms of Schizophrenia in Post-menopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Hospital Sant Joan de Deu (Other); Parc Sanitari Sant Joan de Déu (Other); Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FSJD-RAL-2010
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia in Post Menopausal Women
Keywords: schizophrenia; negative schizophrenia; schizophrenia in post-menopausal women; schizophrenia in women; ralixifene; raloxifen; raloxifeno; negative symptoms of schizophrenia; negative symptoms in schizophrenia; schizophrenia symptoms; negative symptoms of psychosis
MeSH Terms: conditions — Schizophrenia | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raloxifene hydrochloride 60 mg (Experimental): Patients fulfilling inclusion criteria and those giving the general informed consent for the study will be randomly allocated to one of the two groups in the trial (placebo or raloxifene) in a 1:1 proportion and in blocks of 4 patients, using the random number tables designed for this purpose.
  The dose of raloxifene hydrochloride administered will be 60 mg/day. Both placebo and the raloxifene will be administered over 6 months. Patients will take one single daily dose administered in the morning. Both drugs will be given orally in capsule form. The medication of each of the treatment groups (lactose as placebo, raloxifene) will be introduced into dark green gelatin capsules to guarantee the blinding.
  Interventions: Drug: Raloxifene
- Lactosa (placebo) (Placebo Comparator): Patients fulfilling inclusion criteria and those giving the general informed consent for the study will be randomly allocated to one of the two groups in the trial (placebo or raloxifene) in a 1:1 proportion and in blocks of 4 patients, using the random number tables designed for this purpose.
  The dose of raloxifene hydrochloride administered will be 60 mg/day. Both placebo and the raloxifene will be administered over 6 months. Patients will take one single daily dose administered in the morning. Both drugs will be given orally in capsule form. The medication of each of the treatment groups (lactose as placebo, raloxifene) will be introduced into dark green gelatin capsules to guarantee the blinding.
  Interventions: Drug: Lactosa (placebo arm)

INTERVENTIONS:
Drug: Raloxifene — The dose of raloxifene hydrochloride administered will be 60 mg/day. Both placebo and the raloxifene will be administered over 6 months. Patients will take one single daily dose administered in the morning. Drug will be given orally in capsule form.
  Other Names: Raloxifene hydrochloride 60 mg, Laboratory Esteve.
  Arms: Raloxifene hydrochloride 60 mg
Drug: Lactosa (placebo arm) — Both placebo and the raloxifene will be administered over 6 months. Patients will take one single daily dose administered in the morning. Drug will be given orally in capsule form.
  Other Names: Lactosa
  Arms: Lactosa (placebo)

SUMMARY:
The efficacy of raloxifene versus placebo was compared over a six-month period, as an adjuvant treatment of the negative symptoms of schizophrenia in a group of 80 post-menopausal women. The aim of the study is to analyze whether raloxifene has an effect on the positive and negative symptoms of schizophrenia, and on psychopathological symptoms in general, and on social and neuropsychological functioning, and to study the influence of genetic polymorphisms in treatment response.

DETAILED DESCRIPTION:
Several studies have found gender-related differences in the epidemiology, clinical presentation, clinical course and response to treatment of schizophrenic disorder(1,2). Findings relating to a lower frequency of schizophrenia in women, its later onset and less severe clinical course(3,4), have led to the appearance of the "estrogen hypothesis" of schizophrenia, which postulates that estrogen has a protective effect in women susceptible to this disease(5).

The estrogen hypothesis in relation to schizophrenia is based on several studies that showed that estrogen levels are significantly lower in schizophrenic women than in healthy women,(6) and that outbreaks or onset of the disease tend to coincide with stages of the menstrual cycle in which estrogen levels are the lowest(7,8).

Studies on experimental animals have shown that estrogen has a modulating effect on the brain dopaminergic system(9,10) and that it also affects serotoninergic activity(11). Estrogens also enhance neuronal regeneration and block mechanisms of neuronal death(12).

The discovery that estrogen has a modulatory effect on the dopaminergic system has encouraged some researchers to study the therapeutic use of estrogen in schizophrenic patients. Several double-blind clinical trials have shown that estrogens are effective at improving psychotic symptoms(13-15). These last studies analyzed the efficacy of estrogens after one and two months, and mainly in relation to positive symptoms, in patients with the acute illness. However, in older patients it is the severity of the negative, rather than the positive, symptoms that seems to be associated with a poorer cognitive and social function. Moreover, positive symptoms tend to be less severe with age, while negative symptoms tend to persist(16).

Regarding the possible use of estrogens to treat post-menopausal women with schizophrenia, Lindamer et al.,(17) studied the psychopathology of menopausal patients with schizophrenia and found that patients in hormone replacement therapy required lower doses of antipsychotic drugs and presented less negative symptoms, whereas no differences were found in response to treatment in relation to positive symptoms.

The greater frequency of later onset schizophrenia in women than in men seems to be related to the drop in estrogen levels that occurs during the menopause. Häfner et al.(19) found that schizophrenia of late onset was more severe in women than in men, especially in relation to negative symptoms, and these results also appear to support the hypothesis that estrogens act as a protective factor before the menopause.

The use of estrogens as adjuvant therapy in schizophrenia seems promising, although in long-term treatment it can have a potentially negative effect on breast and uterine tissue(20,21). This was the reason we chose raloxifene for our study, which is a selective estrogen receptor modulator (SERM) that can act as a tissue-selective agonist or antagonist. Raloxifene is a first-generation SERM used in the preventive treatment of post-menopausal osteoporosis and does not affect breast or ovarian tissue. (22). It has agonistic effects on the brain(23). Raloxifene seems to influence multiple neurotransmission pathways, including that of seratonin in the frontal cortex, basal and striated ganglia(24), areas of the brain that are commonly affected in schizophrenic patients.

There is some evidence that raloxifene can be useful in the treatment of some mental disorders in post-menopausal women(25,26). Recently, Kulkarni et al.(27) have reported preliminary data that also seem to support a role for raloxifene in schizophrenic patients.

Our team conducted a 12-week, randomized, double-blind, placebo-controlled clinical trial funded by the Stanley Foundation, to assess the value of 60 mg of raloxifene as adjuvant treatment for the negative symptoms, and other psychotic symptoms, in post-menopausal women. In our study on 33 patients, we found that women in the raloxifene group showed a greater improvement in both positive and negative symptoms, and also in general psychopathological symptoms, than women who had only received antipsychotic medication(28).

Since part of Raloxifene's mechanism of action involves activating the estrogenic receptors, some studies have explored the possibility that polymorphisms in these alfa (ESR1) or beta (ESR2) estrogenic receptor genes can modify the effects of treatment with raloxifene(29-31). Several pharmacogenomic studies have reported that single nucleotide polymorphisms (SNPs) in these genes, affect raloxifene treatment in relation to its endothelial function(29), cholesterol levels(30) and bone mineral density(31). Nevertheless, no studies have assessed whether these SNPs of ESR1 or ESR2 can influence raloxifene's effects in the brain. Based on the positive results of our preliminary study, we have designed a longer clinical trial with the same dose of raloxifene that had been effective in the first study. We aim to include in this 6-month placebo-controlled, randomized, double-blind clinical trial a larger number of post-menopausal women with schizophrenia, and improve the clinical assessments by using a larger battery of psychometric tests in areas of social functioning and neuropsychological performance. Genotypic studies will be conducted of the 4 SNPs in the ESR1 (rs9340799, rs2234693, rs1801132) and ESR2 (rs1256049) genes, to control the effects of patients' genotypes on response to treatment.

DESCRIPTION OF THE TARGET POPULATION

The sample includes post-menopausal women diagnosed with schizophrenia according to DSM-IV-TR criteria.

Post-menopause is defined as 1) aged over 45 years with a minimum of one year of amenorrhea and FSH levels higher than 20 UI/L or 2) aged over 50 years old with at least one year of amenorrhea.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of schizophrenia according to DSM-IV TR criteria.
2. Postmenopausal patients. Post-menopausal is defined as 1) aged over 45 years with at least one year of amenorrhea and levels of FSH over 20 UI/L or 2) aged over 50 years with at least one year of amenorrhea.
3. Patients who have been taking a stable dose of antispsychotic medication for at least the 30 days before the start of the study.
4. The presence of significant negative symptoms (defined as one or more negative symptoms with a severity of over 4 on the PANSS scale).
5. General written informed consent by patients or their legal representative.
6. For the genotypic study, a specific informed consent signed by the patients or legal representative is required.

Exclusion criteria:

1. A diagnosis of substance abuse/dependence in the previous 6 months.
2. Mental retardation
3. A diagnosis of major depression (according to DSM-IV TR criteria).
4. Endocrine alterations related to sexual hormones, liver insufficiency including cholestasis, severe renal insufficiency.
5. History or current condition of thromboembolism, breast cancer, abnormal uterine bleeding or stroke.
6. Patients in hormone replacement therapy.
7. Known allergy or hypersensitivity to the active ingredient of the investigational drug, or to any of its excipients or lactose.
8. To be receiving treatment in another clinical trial.
9. To present any severe concomitant disease that in the researcher's opinion can compromise completion of the study or affect the patient's tolerance to this treatment.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of raloxifene (SERM - Selective Estrogen Receptor Modulator) as an adjuvant of antipsychotic treatment in the management of negative symptoms of schizophrenia in post-menopausal women. | Change in score on the negative subscale of the PANSS from baseline to final assessment at week 24
  The primary variable of efficacy will correspond to the change in score on the negative subscale of the PANSS from the start of treatment to the final assessment at 24 weeks. Patients will be considered to respond to treatment if the score in the negative subscale is at least 20% lower than at the start of treatment.

SECONDARY OUTCOMES:
To assess the efficacy of raloxifene as an adjuvant of antipsychotic treatment in the management of global symptoms of schizophrenia in postmenopausal women. | From baseline to week 24 (measurements at Baseline, weeks 4, 12, 24)
  The results from different scales or test will be measured: at baseline,week 4,12 y 24 for scales (PANSS, SANS, CGI, GAF, CDSS -Calgary, LSP, SIMPSON, UKU, DAS-sv) and at baseline, week 12 and 24 for neuropsychological test (TAVEC, CPT, TMT, STROOP, FAS, WAIS sub-tests).
To assess the efficacy of raloxifene as an adjuvant of antipsychotic treatment in the global functioning of postmenopausal women with schizophrenia. | From baseline to week 24 (measurements at Baseline, weeks 4, 12, 24)
  The results from different scales or test will be measured: at baseline,week 4,12 y 24 for scales (PANSS, SANS, CGI, GAF, CDSS -Calgary, LSP, SIMPSON, UKU, DAS-sv) and at baseline, week 12 and 24 for neuropsychological test (TAVEC, CPT, TMT, STROOP, FAS, WAIS sub-tests).
To assess the efficacy of raloxifene as an adjuvant of antipsychotic treatment in the neuropsychological functioning of post-menopausal women with schizophrenia | From baseline to week 24 (measurements at Baseline, week 12, week 24)
  The results from different test will be measured at weeks, baseline, 12 and 24 for neuropsychological test (TAVEC, CPT, TMT, STROOP, FAS, WAIS sub-tests).
To control response to treatment as a function of genetic variants in the form of SNP (Single Nucleotide Polymorphisms) that patients present in the alfa (ESR1) and beta (ESR2) estrogenic receptor genes. | Blood sample collected at Baseline visit
  Analysis will be done for patients who consented by the Informed Consent Form. The analysis will be carried out by centralized laboratory (Biobanc Institut d´Investigació Sanitària Pere Virgili; Reus, Spain) once all samples will be collected. In the meantime, the samples will be kept frozen at 4oC.
To assess the safety of the medication used in this patient population. | From Baseline to week 24
  Safety will be assessed during the study by the vigilance of the AEs, SAEs, AR, SARs at each visit. Blood analysis (hemo/chem) will be done at Baseline and at the end (week 24), and clinical scales will be measured at Baseline, week 4,12 y 24 (PANSS, SANS, CGI, GAF, CDSS -Calgary, LSP, SIMPSON, UKU, DAS-sv)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Usall, PhMD, Principal Investigator — Parc Sanitari Sant Joan de Déu; Javier Labad Arias, PhMD, Principal Investigator — Hospital Psiquiàtric Institut Pere Mata de Reus; Gemma García-Parés, PhMD, Principal Investigator — Corporació Sanitária Parc Taulí
Locations (3):
- Spain (3):
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat, Barcelona
  - Hospital Psiquiàtric Institut Pere Mata, Reus, Tarragona

REFERENCES:
- [Background] Leung A, Chue P. Sex differences in schizophrenia, a review of the literature. Acta Psychiatr Scand Suppl. 2000;401:3-38. doi: 10.1111/j.0065-1591.2000.0ap25.x. PMID 10887978
- [Background] Hafner H. Gender differences in schizophrenia. Psychoneuroendocrinology. 2003 Apr;28 Suppl 2:17-54. doi: 10.1016/s0306-4530(02)00125-7. PMID 12650680
- [Background] Jablensky A, Sartorius N, Ernberg G, Anker M, Korten A, Cooper JE, Day R, Bertelsen A. Schizophrenia: manifestations, incidence and course in different cultures. A World Health Organization ten-country study. Psychol Med Monogr Suppl. 1992;20:1-97. doi: 10.1017/s0264180100000904. No abstract available. PMID 1565705
- [Background] Usall J, Busquets E, Araya S, Ochoa S, Gost A. [Gender differences in schizophrenia. A literature review]. Actas Esp Psiquiatr. 2000 May-Jun;28(3):178-85. Spanish. PMID 11000700
- [Background] Seeman MV, Lang M. The role of estrogens in schizophrenia gender differences. Schizophr Bull. 1990;16(2):185-94. doi: 10.1093/schbul/16.2.185. PMID 2197713
- [Background] Riecher-Rossler A, Hafner H, Stumbaum M, Maurer K, Schmidt R. Can estradiol modulate schizophrenic symptomatology? Schizophr Bull. 1994;20(1):203-14. doi: 10.1093/schbul/20.1.203. PMID 8197416
- [Background] Riecher-Rössler A, Häfner H, Maurer K, Stummbaum M, Schmitd R. Schizophrenia symptomatology varies with serum estradiol levels during menstrual cycle. Schizophrenia Research 1992; 6: 114-115.
- [Background] Huber TJ, Rollnik J, Wilhelms J, von zur Muhlen A, Emrich HM, Schneider U. Estradiol levels in psychotic disorders. Psychoneuroendocrinology. 2001 Jan;26(1):27-35. doi: 10.1016/s0306-4530(00)00034-2. PMID 11070332
- [Background] Di Paolo T, Bedard F, Bedard PJ. Influence of gonadal steroids on human and monkey cerebrospinal fluid homovanillic acid concentrations. Clin Neuropharmacol. 1989 Feb;12(1):60-6. doi: 10.1097/00002826-198902000-00008. PMID 2469538
- [Background] Hafner H, Behrens S, De Vry J, Gattaz WF. An animal model for the effects of estradiol on dopamine-mediated behavior: implications for sex differences in schizophrenia. Psychiatry Res. 1991 Aug;38(2):125-34. doi: 10.1016/0165-1781(91)90038-q. PMID 1754627
- [Background] Moses EL, Drevets WC, Smith G, Mathis CA, Kalro BN, Butters MA, Leondires MP, Greer PJ, Lopresti B, Loucks TL, Berga SL. Effects of estradiol and progesterone administration on human serotonin 2A receptor binding: a PET study. Biol Psychiatry. 2000 Oct 15;48(8):854-60. doi: 10.1016/s0006-3223(00)00967-7. PMID 11063980
- [Background] DonCarlos LL, Azcoitia I, Garcia-Segura LM. Neuroprotective actions of selective estrogen receptor modulators. Psychoneuroendocrinology. 2009 Dec;34 Suppl 1:S113-22. doi: 10.1016/j.psyneuen.2009.04.012. PMID 19447561
- [Background] Kulkarni J, Riedel A, de Castella AR, Fitzgerald PB, Rolfe TJ, Taffe J, Burger H. Estrogen - a potential treatment for schizophrenia. Schizophr Res. 2001 Mar 1;48(1):137-44. doi: 10.1016/s0920-9964(00)00088-8. PMID 11278160
- [Background] Akhondzadeh S, Nejatisafa AA, Amini H, Mohammadi MR, Larijani B, Kashani L, Raisi F, Kamalipour A. Adjunctive estrogen treatment in women with chronic schizophrenia: a double-blind, randomized, and placebo-controlled trial. Prog Neuropsychopharmacol Biol Psychiatry. 2003 Sep;27(6):1007-12. doi: 10.1016/S0278-5846(03)00161-1. PMID 14499318
- [Background] Kulkarni J, de Castella A, Fitzgerald PB, Gurvich CT, Bailey M, Bartholomeusz C, Burger H. Estrogen in severe mental illness: a potential new treatment approach. Arch Gen Psychiatry. 2008 Aug;65(8):955-60. doi: 10.1001/archpsyc.65.8.955. PMID 18678800
- [Background] Bottlender R, Jager M, Groll C, Strauss A, Moller HJ. Deficit states in schizophrenia and their association with the length of illness and gender. Eur Arch Psychiatry Clin Neurosci. 2001 Dec;251(6):272-8. doi: 10.1007/pl00007545. PMID 11881841
- [Background] Lindamer LA, Buse DC, Lohr JB, Jeste DV. Hormone replacement therapy in postmenopausal women with schizophrenia: positive effect on negative symptoms? Biol Psychiatry. 2001 Jan 1;49(1):47-51. doi: 10.1016/s0006-3223(00)00995-1. PMID 11163779
- [Background] Castle D, Sham P, Murray R. Differences in distribution of ages of onset in males and females with schizophrenia. Schizophr Res. 1998 Oct 9;33(3):179-83. doi: 10.1016/s0920-9964(98)00070-x. PMID 9789910
- [Background] Häfner H. Gender differences in first-episode of schizophrenia. In Frank ed, gender and its effects in Psychopathology. American Psychiatric Press, Washington 2000
- [Background] Chlebowski RT, Kuller LH, Prentice RL, Stefanick ML, Manson JE, Gass M, Aragaki AK, Ockene JK, Lane DS, Sarto GE, Rajkovic A, Schenken R, Hendrix SL, Ravdin PM, Rohan TE, Yasmeen S, Anderson G; WHI Investigators. Breast cancer after use of estrogen plus progestin in postmenopausal women. N Engl J Med. 2009 Feb 5;360(6):573-87. doi: 10.1056/NEJMoa0807684. PMID 19196674
- [Background] MacGregor JI, Jordan VC. Basic guide to the mechanisms of antiestrogen action. Pharmacol Rev. 1998 Jun;50(2):151-96. PMID 9647865
- [Background] Huang Y, Huang YL, Lai B, Zheng P, Zhu YC, Yao T. Raloxifene acutely reduces glutamate-induced intracellular calcium increase in cultured rat cortical neurons via inhibition of high-voltage-activated calcium current. Neuroscience. 2007 Jun 29;147(2):334-41. doi: 10.1016/j.neuroscience.2007.04.037. Epub 2007 Jun 1. PMID 17543470
- [Background] Littleton-Kearney MT, Ostrowski NL, Cox DA, Rossberg MI, Hurn PD. Selective estrogen receptor modulators: tissue actions and potential for CNS protection. CNS Drug Rev. 2002 Fall;8(3):309-30. doi: 10.1111/j.1527-3458.2002.tb00230.x. PMID 12353060
- [Background] Jarkova NB, Martenyi F, Masanauskaite D, Walls EL, Smetnik VP, Pavo I. Mood effect of raloxifene in postmenopausal women. Maturitas. 2002 May 20;42(1):71-5. doi: 10.1016/s0378-5122(01)00303-6. PMID 12020982
- [Background] Wong J, Seeman MV, Shapiro H. Case report: raloxifene in postmenopausal women with psychosis: preliminary findings. Am J Geriatr Psychiatry. 2003 Nov-Dec;11(6):697-8. doi: 10.1176/appi.ajgp.11.6.697. No abstract available. PMID 14609815
- [Background] Kulkarni J, Gurvich C, Lee SJ, Gilbert H, Gavrilidis E, de Castella A, Berk M, Dodd S, Fitzgerald PB, Davis SR. Piloting the effective therapeutic dose of adjunctive selective estrogen receptor modulator treatment in postmenopausal women with schizophrenia. Psychoneuroendocrinology. 2010 Sep;35(8):1142-7. doi: 10.1016/j.psyneuen.2010.01.014. Epub 2010 Feb 19. PMID 20171784
- [Background] Usall J, Huerta-Ramos E, Iniesta R, Cobo J, Araya S, Roca M, Serrano-Blanco A, Teba F, Ochoa S. Raloxifene as an adjunctive treatment for postmenopausal women with schizophrenia: a double-blind, randomized, placebo-controlled trial. J Clin Psychiatry. 2011 Nov;72(11):1552-7. doi: 10.4088/JCP.10m06610. Epub 2011 Aug 23. PMID 21903021
- [Background] Zavratnik A, Zegura B, Marc J, Prezelj J, Pfeifer M. XbaI polymorphism of the estrogen receptor alpha gene influences the effect of raloxifene on the endothelial function. Maturitas. 2010 Sep;67(1):84-90. doi: 10.1016/j.maturitas.2010.05.011. Epub 2010 Jul 6. PMID 20609538
- [Background] Zavratnik A, Prezelj J, Kocijancic A, Marc J. Exonic, but not intronic polymorphisms of ESR1 gene might influence the hypolipemic effect of raloxifene. J Steroid Biochem Mol Biol. 2007 Apr;104(1-2):22-6. doi: 10.1016/j.jsbmb.2006.10.009. Epub 2007 Mar 12. PMID 17350824
- [Background] Zhang ZL, He JW, Qin YJ, Huang QR, Liu YJ, Hu YQ, Li M. Association of bone metabolism related genes polymorphisms with the effect of raloxifene hydrochloride on bone mineral density and bone turnover markers in postmenopausal women with osteoporosis. Zhonghua Yi Xue Yi Chuan Xue Za Zhi. 2006 Apr;23(2):129-33. PMID 16604479
- [Result] Chua WL, de Izquierdo SA, Kulkarni J, Mortimer A. Estrogen for schizophrenia. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD004719. doi: 10.1002/14651858.CD004719.pub2. PMID 16235377
- [Derived] Huerta-Ramos E, Labad J, Cobo J, Nunez C, Creus M, Garcia-Pares G, Cuadras D, Franco J, Miquel E, Reyes JC, Marco-Garcia S; RALOPSYCAT Group; Usall J. Effects of raloxifene on cognition in postmenopausal women with schizophrenia: a 24-week double-blind, randomized, parallel, placebo-controlled trial. Eur Arch Psychiatry Clin Neurosci. 2020 Sep;270(6):729-737. doi: 10.1007/s00406-019-01079-w. Epub 2019 Nov 14. PMID 31728631
- [Derived] Usall J, Huerta-Ramos E, Labad J, Cobo J, Nunez C, Creus M, Pares GG, Cuadras D, Franco J, Miquel E, Reyes JC, Roca M; RALOPSYCAT Group. Raloxifene as an Adjunctive Treatment for Postmenopausal Women With Schizophrenia: A 24-Week Double-Blind, Randomized, Parallel, Placebo-Controlled Trial. Schizophr Bull. 2016 Mar;42(2):309-17. doi: 10.1093/schbul/sbv149. Epub 2015 Nov 20. PMID 26591005